CLINICAL TRIAL: NCT01786148
Title: An Audio Music Self-Management Program to Improve ART Adherence in Rural GA
Brief Title: Music for Health Project
Acronym: MFH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Marcia McDonnell Holstad, DSN, FNP-BC, Associate Professor, Emory University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00055077; 1R01NR012923 (NIH)
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Results first posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV/AIDS; Adherence; Self-management; Antiretroviral therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational music mobile app (Active Comparator): A prerecorded program of songs on various topics in a mobile phone application (app). It is designed to provide education about non-health related topics and will be equivalent in length to the intervention app.
  Interventions: Behavioral: mobile phone application
- Live Network mobile phone App (Experimental): The LN is a prerecorded mobile phone application (app). It employs a radio talk show format in which a Disc Jockey entertains HIV medication-, adherence-, and self-management-related questions and comments from callers and poses them to expert care providers, whose responses to these questions are augmented by songs that shed additional light on these issues.
  Interventions: Behavioral: mobile phone application

INTERVENTIONS:
Behavioral: mobile phone application

SUMMARY:
The overall goal of this project is to use technology to improve adherence to antiretroviral therapy (ART)and increase access to ART adherence care for those HIV+ persons living in rural areas. The LIVE Network audio music program mobile application (app) is innovative, practical, portable, and could be rapidly scaled up to address the adherence self-management needs of rural groups nationwide. If successful, the impact on HIV care will be immense and could transform the delivery of HIV self-management and adherence education by overcoming barriers of geographic isolation, transportation, stigma and confidentiality in this vulnerable group.

DETAILED DESCRIPTION:
The project has two primary aims and one exploratory aim. 1.0 Revise and adapt the Live Network (LN) program and manual for rural persons living with HIV/AIDS (PLWHA) and develop into a mobile application.

2.0 Conduct a randomized controlled trial to test the efficacy of the program. When compared with an educational music control condition at 3, 6, and 9 months post-baseline, those randomized to the LN will have: H1: Significantly higher mean antiretroviral therapy (ART) adherence rates (measured by pill counts, self report).

H2: Significantly higher mean levels of ART drug levels in hair sample analyses.

H3: Significantly better clinical indicators: higher mean CD4 lymphocyte counts and percents, a larger proportion achieving virologic suppression (proportion with HIV RNA PCR <50 copies/ml), and smaller proportion with evidence of drug resistance, all as measured by medical record review.

3.0 Explore: a) the effects of LN on symptoms and symptom management; b) the roles of self-efficacy, outcome expectancies, and personal goal setting as mediators, and depression and health literacy as moderators of adherence.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ individuals initiating ART for the first time (except women who may have had ART during pregnancy); or HIV+ individuals changing ART regimen within the past 3 months due to side effects or virologic resistance; or HIV+ individuals with a detectable viral load ≥ 40copies/ml; or HIV+ individuals on ART medication
* English speaking
* Willing to complete 4 assessments
* Willing to complete monthly, unannounced pill counts
* Willing to allow collection of hair samples
* Willing to be randomly assigned to either condition
* Willing to participate in study activities that include using smart phone and mobile app

Exclusion Criteria:

* Have a history of bilateral hearing loss (health care provider diagnosed or self-identified)
* Homeless
* Have a cognitive impairment (inability to comprehend the informed consent)
* Display psychotic symptoms, as determined by the Brief Symptom Inventory (BSI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2014-06; Primary Completion 2017-04-19 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia M Holstad, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the trial starting in June 2014 and randomized either to Educational music mobile app or to the Live Network mobile phone app
Groups:
- Educational Music Mobile App: A prerecorded program of songs on various topics in a mobile phone application (app). It is designed to provide education about non-health related topics and will be equivalent in length to the intervention app.
  mobile phone application
- Live Network Mobile Phone App: The LN is a prerecorded mobile phone application (app). It employs a radio talk show format in which a Disc Jockey entertains HIV medication-, adherence-, and self-management-related questions and comments from callers and poses them to expert care providers, whose responses to these questions are augmented by songs that shed additional light on these issues.
  mobile phone application
Period: Overall Study
Arm/Group | Educational Music Mobile App | Live Network Mobile Phone App
Started | 77 | 72
Completed | 55 | 50
Not Completed | 22 | 22
Not completed — Lost to Follow-up | 21 | 13
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 7
Not completed — Incarceration | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Educational Music Mobile App | Live Network Mobile Phone App | Total
Number analyzed (Participants) | 77 | 72 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (11.6) | 37.3 (11.1) | 39.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 51
  Male | 49 | 49 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 61 | 54 | 115
  White | 8 | 15 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 2 | 9
Consider Yourself to be [Count of Participants; unit: Participants]
  Straight/Heterosexual | 42 | 29 | 71
  Gay/Homosexual | 28 | 27 | 55
  Bisexual | 5 | 12 | 17
  None of the above | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Antiretroviral Therapy (ART) Adherence Rates
Description: Adherence rate was measured with the Antiretroviral General Adherence Scale (AGAS) which measures the general ease and ability to take one's medication as prescribed in the past 30 days. It includes 5 items scored 1 to 6, with the possible scores for this instrument ranging from 5 to 30, and higher scores reflect better adherence.
Time Frame: Baseline, 3 months post-baseline, 6 months post-baseline and 9 months post-baseline
Population: Population included only subjects that were able to complete the Antiretroviral General Adherence Scale (AGAS) which measures the general ease and ability to take one's medication as prescribed in the past 30 days. The possible scores for this instrument range from 5 to 30, and higher scores reflect better adherence.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Educational Music Mobile App | Live Network Mobile Phone App
Number analyzed (Participants) | 64 | 60
score on a scale
  Baseline | 27.04 (4.23) | 26.25 (5.18)
  3 months | 26.14 (4.81) | 26.48 (5.39)
  6 months | 26.60 (5.48) | 27.81 (3.90)
  9 months | 26.45 (5.90) | 26.38 (5.99)

2. Secondary Outcome: Change in Antiretroviral (ART) Drug Levels in Hair Sample Analyses.
Description: No data available due to inability of the lab to accurately extract drug from hair.
Time Frame: 3, 6, and 9 months post-baseline
Population: Data were not collected.
Arm/Group | Educational Music Mobile App | Live Network Mobile Phone App
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Clinical Indicator: Change in Mean CD4 Percentage
Description: CD4 count is a test that measures the number of CD4 cells in your blood. CD4 cells, also known as T cell lymphocytes, are white blood cells that fight infection and play an important role in your immune system. A CD4 count is used to check the health of the immune system in people infected with HIV (human immunodeficiency virus). The count measures the number of CD4 cells in a small sample of blood. The percent of CD4 cells measure the percentage of all lymphocytes that are CD4 cells. The study assesses the percentage of CD4 lymphocytes over time.
Time Frame: Baseline, 3 months post-intervention, 6 months post-intervention, 9 months post-intervention, 9 to 12 months post-intervention
Population: Population includes participants with a valid CD4 sample analyzed.
Measure: Mean (Standard Deviation); unit: percentage of CD4
Arm/Group | Educational Music Mobile App | Live Network Mobile Phone App
Number analyzed (Participants) | 60 | 51
percentage of CD4
  Baseline: number analyzed (Participants) | 52 | 50
  Baseline | 21.87 (12.66) | 26.07 (14.26)
  3 months post-intervention: number analyzed (Participants) | 60 | 43
  3 months post-intervention | 21.68 (12.37) | 25.91 (12.32)
  6 months post-intervention: number analyzed (Participants) | 48 | 51
  6 months post-intervention | 27.08 (12.90) | 26.23 (13.27)
  9 months post-intervention: number analyzed (Participants) | 37 | 40
  9 months post-intervention | 26.13 (11.92) | 24.08 (14.08)
  9 to 12 months post-intervention: number analyzed (Participants) | 32 | 32
  9 to 12 months post-intervention | 24.80 (11.40) | 26.39 (10.49)

4. Secondary Outcome: Clinical Indicator: Number of Participants With Non-detectable Viral Load
Description: Change in number of participants with viral load presented as number of copies if <50 copies versus ≥ 50 copies. Subjects were coded as having non-detectable viral loads if the "load" was < 50 copies. The analyses performed reflects the number of subjects with non-detectable load (<50) at Baseline, 3 months post-intervention, 6 months post-intervention, 9 months post-intervention, 9 to 12 months post-intervention.
Time Frame: as for outcome 3
Population: Only number of participants with available lab tests are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Educational Music Mobile App | Live Network Mobile Phone App
Number analyzed (Participants) | 64 | 56
Participants
  Baseline: number analyzed (Participants) | 62 | 56
  Baseline | 25 | 21
  3 months post-intervention: number analyzed (Participants) | 64 | 47
  3 months post-intervention | 49 | 35
  6 months post-intervention: number analyzed (Participants) | 48 | 47
  6 months post-intervention | 40 | 38
  9 months post-intervention: number analyzed (Participants) | 36 | 41
  9 months post-intervention | 27 | 33
  9 to 12 months post-intervention: number analyzed (Participants) | 34 | 32
  9 to 12 months post-intervention | 26 | 27

ADVERSE EVENTS:
Time Frame: 9 months post-baseline
Groups:
- Live Network Mobile Phone App: The Live Network (LN) is a prerecorded mobile phone application (app). It employs a radio talk show format in which a Disc Jockey entertains HIV medication-, adherence-, and self-management-related questions and comments from callers and poses them to expert care providers, whose responses to these questions are augmented by songs that shed additional light on these issues.
  mobile phone application
Arm/Group | Educational Music Mobile App | Live Network Mobile Phone App
All-Cause Mortality (participants affected / at risk) | 0/77 | 1/72
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/72
Other Adverse Events (participants affected / at risk) | 0/77 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT01786148/Prot_SAP_000.pdf